CLINICAL TRIAL: NCT05988047
Title: Analysis of CMTM6 Expression in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Professor, University of Freiburg
Other Study IDs: CMTM6_AML
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AML: Peripheral blood will be taken at the timepoint of primary diagnosis and analyzed for CMTM6 expression and T cell activation
- Healthy controls: Peripheral blood will be taken analyzed for CMTM6 expression and T cell activation

SUMMARY:
In this study, we aim to investigate the expression of CKLF like MARVEL transmembrane domain containing 6 (CMTM6) in leukemia cells of patients with acute myeloid leukemia (AML). We will use peripheral blood samples and assess CMTM6 expression by flow cytometry and Western Blot.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* primary diagnosis of acute myeloid leukemia
* diagnosis results available
* written informed consent
* ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* lack of informed consent

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with AML at primary diagnosis ≥ 18 years of age
  or
  healthy probands ≥ 18 years of age
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
CMTM6 expression (FC) | At primary diagnosis
  CMTM6 expression on blasts/monocytes will be measured by flow cytometry
T cell activation (FC) | At primary diagnosis
  T cell activation and cytokine production will be measured by flow cytometry

SECONDARY OUTCOMES:
CMTM6 expression (WB) | At primary diagnosis
  CMTM6 expression on blasts/monocytes will be measured by Western blot

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center- University of Freiburg, Freiburg im Breisgau, CA, Germany

IPD SHARING:
Plan to Share IPD: No